CLINICAL TRIAL: NCT01917110
Title: Efficacy and Safety of MiSight ® Contact Lenses in Reducing the Progression of Childhood Myopia, Not Pathological, Aged 8-12 Years Randomized Clinical Trial.
Brief Title: Efficacy and Safety of MiSight ® Contact Lenses in Reducing the Progression of Childhood Myopia.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CooperVision, Inc. (Industry)
Responsible Party: Sponsor
Organization: CooperVision International Limited (CVIL) (Industry)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P2013/05
Record Dates: First submitted 2013-08-02; First posted 2013-08-06 (Estimated); Last update posted 2020-08-03 (Actual); Status verified 2020-07

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia | interventions — Eyeglasses

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- omafilcon A (Experimental): Contact Lens Group
  Interventions: Device: omafilcon A
- Spectacle Group (Active Comparator): Prescription at Baseline
  Interventions: Device: Spectacle

INTERVENTIONS:
Device: omafilcon A
  Arms: omafilcon A
Device: Spectacle
  Arms: Spectacle Group

SUMMARY:
The purpose of the study is to quantify the effectiveness of CooperVision MiSight® (omafilcon A) soft (hydrophilic) contact lens in slowing the rate of progression of juvenile-onset myopia.

DETAILED DESCRIPTION:
Subjects in two parallel groups were randomized and assigned to either the study contact lens (omafilcon a) or single vision spectacles.

ELIGIBILITY:
Inclusion Criteria:

* Prior to being considered eligible to participate in this study, each subject MUST:

  1. Be between 8 and 12 years of age inclusive at the baseline examination.
  2. Have:

     1. read the Informed Assent,
     2. been given an explanation of the Informed Assent,
     3. indicated an understanding of the Informed Assent and
     4. signed the Informed Assent Form.
  3. Have their parent or legal guardian:

     1. read the Informed Consent,
     2. been given an explanation of the Informed Consent,
     3. indicated an understanding of the Informed Consent and
     4. signed the Informed Consent Form.
  4. Along with their parent or guardian, be capable of comprehending the nature of the study, and be willing and able to adhere to the instructions set forth in this protocol.
  5. Along with their parent or guardian, agree to maintain the visit schedule and be able to keep all appointments as specified in the study protocol for the duration of the study
  6. Agree to accept either the control or test lens as assigned by the randomisation scheme.
  7. Agree to wear the assigned contact lenses for the duration of the 2 year study and to inform the study investigator if this schedule is interrupted. (Wearing time may be modified by the study staff for health reasons.)
  8. Possess wearable and visually functional eyeglasses.
  9. Be in good general health, based on his/her and parent's/guardian's knowledge.
  10. Have best-corrected visual acuity by manifest refraction of +0.10 logMAR (20/25 Snellen equivalent) or better in each eye.
  11. Meet the following refractive criteria determined by cycloplegic autorefraction at baseline:

      1. Spherical Equivalent Refractive Error (SERE): between -0.75 and -4.00 D inclusive.
      2. Astigmatism: < -0.75 D
      3. Anisometropia: < 1.00D

Exclusion Criteria:

* Subjects may not be considered eligible if ANY of the following apply:

  1. Subject has previously or recently worn soft or rigid gas permeable contact lenses, including orthokeratology lenses.
  2. Subject appears to exhibit poor personal hygiene (that in the investigator's opinion might prevent safe contact lens wear).
  3. Subject is currently or prior to this study has been an active participant in another clinical study.
  4. Parent / guardian or close relative is a member, of the office staff, including the investigator(s).
  5. Current or prior use of bifocals, progressive addition lenses, atropine, pirenzepine or ANY other myopia control treatment.
  6. Subject was born earlier than 30 weeks or weighed less than 1500g (3.3lb) at birth.
  7. Regular use of ocular medications (prescription or over-the-counter), artificial tears, or wetting agents.
  8. Current use of systemic medications which may significantly affect contact lens wear, tear film production, pupil size, accommodation or refractive state. Such as, but not limited to: long term use of nasal decongestants (for example, pseudoephedrine, phenylephrine), antihistamines (for example, chlorpheniramine, diphenhydramine), Prednisolone or Ritalin (methylphenidate).
  9. A known allergy to fluorescein, benoxinate, proparacaine or tropicamide.
  10. A history of corneal hypoesthesia (reduced corneal sensitivity), corneal ulcer, corneal infiltrates, ocular viral or fungal infections or other recurrent ocular infections.
  11. Strabismus by cover test at far (4 m) or near (40 cm) wearing distance correction.
  12. Known ocular or systemic disease such as, but not limited to: anterior uveitis or iritis, episcleritis or scleritis, glaucoma, Sjogren's syndrome, lupus erythematosus, scleroderma, or diabetes.
  13. Any ocular, systemic or neuro-developmental conditions that could influence refractive development. Such as, but not limited to: persistent pupillary membrane, vitreous hemorrhage, cataract, corneal scarring, ptosis eyelid hemangiomas, Marfan's Syndrome, Down's syndrome, Ehler's-Danlos syndrome, Stickler's syndrome, ocular albinism, retinopathy of prematurity.
  14. Keratoconus or an irregular cornea.
  15. Biomicroscope findings that would contraindicate contact lens wear including, but not limited to:

      1. corneal scars within the visual axis
      2. neovascularisation or ghost vessels > 1.5 mm in from the limbus
      3. Any active anterior segment ocular disease that would contraindicate contact lens wear.
      4. giant papillary conjunctivitis of Grade 2 or worse
      5. allergic or seasonal conjunctivitis (if the study investigator believes it could significantly interfere with maintaining the specified contact lens wearing schedule)
      6. clinically significant (Grade 3 or 4) abnormalities of the anterior segment, lids, conjunctiva, sclera or associated structures.
  16. The investigator for any reason considers that it is not in the best interest of the subject to participate in the study.
  17. Have pathological myopia To be eligible to begin the study, a subject must have ALL of the inclusion criteria and NONE of the exclusion criteria present.

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 79 (Actual)
Dates: Start 2013-09-13 (Actual); Primary Completion 2016-06-16 (Actual); Study Completion 2016-06-16 (Actual)

PRIMARY OUTCOMES:
Change in the spherical equivalent refractive error relative to baseline. | Baseline, 1 week, 1 month, 6 months, 12 months, 18 months, 24 months
Change in axial length relative to baseline. | Baseline, 1 week, 1 month, 6 months, 12 months, 18 months, 24 months
Measurement of corneal curvature (keratometry)relative to baseline. | Baseline, 1 week, 1 month, 6 months, 12 months, 18 months, 24 months

SECONDARY OUTCOMES:
Measurement of pupil diameter relative to baseline. | Baseline, 1 week, 1 month, 6 months, 12 months, 18 months, 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Cesar Villa Collar, OD PhD FAAO, Principal Investigator — Departamento de Optica y Optometria de la Universidad Europea de Madrid
Locations (1):
- Departamento de Óptica y Optometría de la Universidad Europea de Madrid, Madrid, Spain

REFERENCES:
- [Derived] Lawrenson JG, Shah R, Huntjens B, Downie LE, Virgili G, Dhakal R, Verkicharla PK, Li D, Mavi S, Kernohan A, Li T, Walline JJ. Interventions for myopia control in children: a living systematic review and network meta-analysis. Cochrane Database Syst Rev. 2023 Feb 16;2(2):CD014758. doi: 10.1002/14651858.CD014758.pub2. PMID 36809645
- [Derived] Lopes-Ferreira D, Ruiz-Pomeda A, Perez-Sanchez B, Queiros A, Villa-Collar C. Ocular and corneal aberrations changes in controlled randomized clinical trial MiSight(R) Assessment Study Spain (MASS). BMC Ophthalmol. 2021 Mar 1;21(1):112. doi: 10.1186/s12886-021-01865-y. PMID 33648464
- [Derived] Ruiz-Pomeda A, Prieto-Garrido FL, Hernandez Verdejo JL, Villa-Collar C. Rebound Effect in the Misight Assessment Study Spain (Mass). Curr Eye Res. 2021 Aug;46(8):1223-1226. doi: 10.1080/02713683.2021.1878227. Epub 2021 Jan 24. PMID 33460537
- [Derived] Ruiz-Pomeda A, Perez-Sanchez B, Canadas P, Prieto-Garrido FL, Gutierrez-Ortega R, Villa-Collar C. Binocular and accommodative function in the controlled randomized clinical trial MiSight(R) Assessment Study Spain (MASS). Graefes Arch Clin Exp Ophthalmol. 2019 Jan;257(1):207-215. doi: 10.1007/s00417-018-4115-5. Epub 2018 Sep 8. PMID 30196481
- [Derived] Ruiz-Pomeda A, Perez-Sanchez B, Valls I, Prieto-Garrido FL, Gutierrez-Ortega R, Villa-Collar C. MiSight Assessment Study Spain (MASS). A 2-year randomized clinical trial. Graefes Arch Clin Exp Ophthalmol. 2018 May;256(5):1011-1021. doi: 10.1007/s00417-018-3906-z. Epub 2018 Feb 3. PMID 29396662